CLINICAL TRIAL: NCT02966756
Title: A Phase 2 Open-Label Study of the Efficacy of Venetoclax in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of Venetoclax in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-728
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Relapsed chronic lymphocytic leukemia (CLL); Refractory chronic lymphocytic leukemia (CLL); 17p deletion; Venetoclax; Leukemia; Lymphoproliferative Disorders; Small Lymphocytic Lymphoma (SLL); Venclexta
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion; Leukemia; Lymphoproliferative Disorders | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Venetoclax (Experimental): Participants with 17p deletion status will receive various doses of venetoclax once daily (QD).
  Interventions: Drug: Venetoclax
- Cohort 2: Venetoclax (Experimental): Participants who have failed a B-Cell Receptor Signaling Pathway Inhibitor (BCRI) therapy and who have also failed, or were unable to receive chemoimmunotherapy (CIT) irrespective of 17p status will receive various doses of venetoclax once daily (QD).
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Tablet; Oral
  Other Names: ABT-199; GDC-0199; Venclexta

SUMMARY:
This is a Phase 2, open-label, multicenter study, evaluating the efficacy of venetoclax in participants with relapsed or refractory Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) either in presence of 17p deletion (Cohort 1) or those who have failed a B-receptor signaling pathway inhibitor (BCRI) therapy and who have also failed, or were unable to receive chemoimmunotherapy (CIT) irrespective of 17p status (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of relapsed or refractory chronic lymphocytic leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) that meets 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (iwCLL) National Cancer Institute-Working Group (NCI-WG) Guidelines and the following:

  * Participant must have an indication for treatment according to the 2008 Modified iwCLL NCI-WG Guidelines.
  * SLL participant must have measurable disease (B-lymphocytosis greater than 5 × 10^9/L or an enlarged lymph node(s) (Longest Diameter (LDi) > 1.5 cm at baseline) or hepatomegaly or splenomegaly due to CLL).
  * SLL participant must have presence of lymphadenopathy and absence of cytopenias caused by a clonal marrow infiltrate.
  * Participant must have relapsed or refractory CLL/SLL after receiving at least one prior line of therapy.
* Participants (in Cohort 1) must have 17p deletion, assessed by a central laboratory.
* Participants (in Cohort 2) must meet both of the following:

  * Relapsed/refractory disease to B-Cell Receptor Signaling Pathway Inhibitor (BCRI) treatment;
  * And either of the following: (a) relapsed/refractory disease to chemoimmunotherapy (CIT), or (b) ineligible to receive CIT, defined as having known 17p deletion or TP53 mutation, or Cumulative Illness Rating Scale (CIRS) >6 or calculated creatinine clearance <70 mL/min, or participants in whom the investigator evaluated that the use of CIT was inappropriate.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
* Participant must have adequate bone marrow function, coagulation profile, renal, and hepatic function, per laboratory reference range at Screening.
* No known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

Exclusion Criteria:

* Participant has undergone an allogeneic stem cell transplant.
* Participant has developed Richter's transformation confirmed by biopsy.
* Participant has prolymphocytic leukemia.
* Participant has active and uncontrolled autoimmune cytopenias (for 2 weeks prior to screening), including autoimmune hemolytic anemia (AIHA) and idiopathic thrombocytopenic purpura (ITP).
* Participant has previously received venetoclax or other BCL-2 inhibitors.
* Participant is known to be positive for Human Immunodeficiency Virus (HIV).
* Participant has received a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Participant has received any of the following within 14 days or 5 half-lives (whichever is shorter) prior to the first dose of venetoclax, or has not recovered to less than Common Toxicity Criteria for Adverse Events (CTCAE) grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

  * Any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy or targeted small molecule agents.
  * Investigational therapy, including targeted small molecule agents.
* Participant has known allergy to both xanthine oxidase inhibitors and rasburicase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Measured up to 2 years after the last participant has enrolled in the study.
  ORR is the proportion of participants with an overall response (complete remission [CR], plus complete remission with incomplete bone marrow recovery [CRi], plus nodular partial remission [nPR], plus partial remission [PR]) per the National Cancer Institute-Working Group (NCI-WG) guidelines as assessed by the Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Measured up to 2 years after the last participant has enrolled into the study.
  CRR is defined as the proportion of subjects who achieved (CR + CRi) per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (iwCLL) NCI-WG criteria.
Duration of Overall Response (DOR) | Measured up to 2 years after the last participant has enrolled into the study.
  DOR is defined as the number of days from the date of first (CR + CRi + nPR + PR) to the earliest disease progression or death
Progression Free Survival (PFS) | Measured up to 5 years after the last participant has enrolled into the study.
  PFS is defined as the number of days from the date of first dose to the date of earliest disease progression (determined by the IRC) or death.
Event Free Survival (EFS) | Measured up to 5 years after the last participant has enrolled into the study.
  EFS is defined as the number of days from the date of first dose to the date of earliest disease progression, death, or start of a new anti-leukemic therapy.
Time to Progression (TTP) | Measured up to 5 years after the last participant has enrolled into the study.
  TTP is defined as the number of days from the date of first dose to the date of earliest disease progression (determined by the IRC).
Time to 50% reduction in absolute lymphocyte count (ALC) | Measured up to 2 years after the last participant has enrolled into the study.
  Time to 50% reduction in ALC is defined as the number of days from the date of first dose to the date when the ALC has reduced to 50% of the baseline value.
Overall Survival (OS) | Measured up to 5 years after the last participant has enrolled into the study.
  OS is defined as number of days from the date of first dose to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (31):
- Australia (3):
  - Concord Repatriation General Hospital /ID# 201261, Concord, New South Wales
  - St George Hospital /ID# 206484, Kogarah, New South Wales
  - Monash Health - Monash Medical Centre /ID# 201263, Clayton, Victoria
- China (21):
  - Anhui Provincial Cancer Hospital /ID# 209458, Hefei, Anhui
  - Peking University People's Hospital /ID# 156575, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 156576, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital /ID# 156579, Fuzhou, Fujian
  - Guangdong Provincial Peoples Hospital /ID# 160509, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 156571, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 159143, Shijiazhuang, Hebei
  - Henan Cancer Hospital /ID# 156573, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College of HUST /ID# 156589, Wuhan, Hubei
  - Xiangya Hospital Central South University /ID# 208913, Changsha, Hunan
  - Jiangsu Province Hospital /ID# 156577, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 156536, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 159142, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 156532, Changchun, Jilin
  - Shandong Provincial Hospital /ID# 156574, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 156572, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 156537, Chengdu, Sichuan
  - The General Hospital of Western Theater Command PLA /ID# 159145, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 157762, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital /ID# 156542, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 156578, Hangzhou, Zhejiang
- New Zealand (2):
  - North Shore Hospital /ID# 204637, Takapuna, Auckland
  - Christchurch Hospital. /ID# 201650, Christchurch, Canterbury
- Taiwan (5):
  - National Taiwan University Hospital /ID# 210733, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 202768, Changhua City, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 202765, Kaohsiung City
  - China Medical University Hospital /ID# 202767, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 203636, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M14-728